CLINICAL TRIAL: NCT02045095
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation Study to Assess the Safety and Tolerability of MLN7243, an Inhibitor of Ubiquitin-Activating Enzyme (UAE), in Adult Patients With Advanced Solid Tumors
Brief Title: A Dose Escalation Study of MLN7243 (TAK-243) in Adult Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C33001; U1111-1203-6359 (Other: WHO)
Record Dates: First submitted 2013-12-18; First posted 2014-01-24 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Drug therapy
MeSH Terms: interventions — TAK-243

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Schedule A: MLN7243 1 mg (Experimental): MLN7243 1 milligram (mg), infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or disease progression (PD) or discontinuation of study for another reason, or until study is stopped.
  Interventions: Drug: MLN7243
- Schedule A: MLN7243 2 mg (Experimental): MLN7243 2 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD, or discontinuation of study for another reason, or until study is stopped.
  Interventions: Drug: MLN7243
- Schedule A: MLN7243 4 mg (Experimental): MLN7243 4 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
  Interventions: Drug: MLN7243
- Schedule A: MLN7243 8 mg (Experimental): MLN7243 8 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
  Interventions: Drug: MLN7243
- Schedule A: MLN7243 12 mg (Experimental): MLN7243 12 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
  Interventions: Drug: MLN7243
- Schedule A: MLN7243 18 mg (Experimental): MLN7243 18 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
  Interventions: Drug: MLN7243
- Schedule A: MLN7243 Homozygous Mutant 4 mg (Experimental): MLN7243 homozygous mutant 4 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
  Interventions: Drug: MLN7243

INTERVENTIONS:
Drug: MLN7243 — Dose escalation stage Schedule A: Intravenous infusion on Days 1, 4, 8, 11 for a 21-day treatment cycle.
  Schedule B: Intravenous infusion on Days 1, 8, 15 for a 28-day treatment cycle.
  Dose expansion stage: MLN7243 will be administered following schedule A (twice-weekly, 21-day dosing) and/or B (once-weekly, 28-day dosing).
  Other Names: TAK-243

SUMMARY:
The purpose of this study is to evaluate safety and tolerability (establish maximum tolerated dose [MTD], inform the recommended phase 2 dose [RP2D], and identify the dose-limiting toxicities [DLTs]) of MLN7243.

DETAILED DESCRIPTION:
This is a single arm Phase I study with multiple dosing cohorts as noted below:

* Schedule A: MLN7243 1 mg
* Schedule A: MLN7243 2 mg
* Schedule A: MLN7243 4 mg
* Schedule A: MLN7243 8 mg
* Schedule A: MLN7243 12 mg
* Schedule A: MLN7243 18 mg
* Schedule A: MLN7243 Homozygous Mutant 4 mg

ELIGIBILITY:
Inclusion Criteria

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

1. Male or female participants 18 years or older.
2. Participants must have a histologically confirmed diagnosis of an advanced, metastatic malignant solid tumor and must have failed or exhausted standard therapies or for which no standard therapy is available.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Participants with adequate hematologic and organ function.
5. All participants must have radiographically detectable tumors with measurable disease as defined by RECIST (version 1.1).
6. Participants undergoing a biopsy procedure must have accessible lesions which are safe to biopsy.
7. Recovered (that is, less than or equal to (<=) Grade 1 toxicity) from the reversible effects of prior antineoplastic therapy, except alopecia.
8. Female participants who are postmenopausal for at least 1 year before the screening visit, surgically sterile, or agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 4 months after the last dose of study drug, or agree to practice true abstinence.

   Male participants who agree to practice effective barrier contraception during the entire study treatment period through 4 months after the last dose of study drug or agree to practice true abstinence.
9. Suitable venous access for the study-required blood sampling including PK sampling.

Exclusion Criteria

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Participants with clinically significant pre-existing cardiac impairment.
2. Participants homozygous for the ABCG2 (BCRP) c.421C greater than (>) 1 A polymorphism will be excluded from the study until the safety of a minimum of the first 3 dose levels has been characterized and the sponsor confirms that such participants can be enrolled at doses that are at least 3-fold lower than the most recently determined safe and tolerable dose among at least 3 dose limiting toxicities (DLT)-evaluable non-homozygous participants.
3. Participants with known active central nervous system (CNS) lesions are excluded. Systemic antineoplastic therapy or investigational agents within 21 days before the first dose of study drug.
4. Radiotherapy within 14 days before the first dose of study drug is not allowed except for limited field radiotherapy for palliative bone pain.
5. For participants where tumor biopsies are required or requested:

   * Any known coagulation abnormalities that would contraindicate the tumor biopsy procedure.
   * Ongoing therapy with any anticoagulant or antiplatelet agents (example, aspirin, clopidogrel [Plavix®], heparin, or warfarin).
6. Major surgery within 28 days before the first dose of MLN7243.
7. Life-threatening illness unrelated to cancer.
8. Any evidence of active infection or antibiotic therapy within 14 days before the first dose of MLN7243.
9. Known human immunodeficiency virus (HIV) positivity or AIDS-related illness, hepatitis B virus, and hepatitis C virus.
10. Participants whose weight is less than (<) 40 kilogram (kg).
11. History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease.
12. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Boston, Massachusetts
  - St Louis, Missouri
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in the United States from 31 January 2014 to 09 November 2016.
Pre-assignment Details: Participants with diagnosis of advanced malignant solid tumors were enrolled in Schedule A of dose escalation phase to receive TAK-243 (MLN7243). The study was terminated prior to start of Schedule B of dose escalation phase and planned expansion because of realignment of the sponsor's pipeline program.
Groups:
- Schedule A: TAK-243 1 mg: TAK-243 (MLN7243) 1 milligram (mg), infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or disease progression (PD) or discontinuation of study for another reason, or until study is stopped.
- Schedule A: TAK-243 2 mg: TAK-243 (MLN7243) 2 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD, or discontinuation of study for another reason, or until study is stopped.
- Schedule A: TAK-243 4 mg: TAK-243 (MLN7243) 4 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
- Schedule A: TAK-243 8 mg: TAK-243 (MLN7243) 8 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
- Schedule A: TAK-243 12 mg: TAK-243 (MLN7243) 12 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
- Schedule A: TAK-243 18 mg: TAK-243 (MLN7243) 18 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
- Schedule A: TAK-243 Homozygous Mutant 4 mg: TAK-243 (MLN7243) homozygous mutant 4 mg, infusion, intravenously over 10-minutes, on Days 1, 4, 8, and 11 followed by 10 days of rest in a 21-day treatment cycle for a maximum of 12 months, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
Period: Overall Study
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Started | 3 | 4 | 4 | 4 | 5 | 8 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 4 | 4 | 5 | 8 | 1
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Progressive Disease | 3 | 3 | 2 | 4 | 2 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of TAK-243.
Groups:
- Schedule A: TAK-243 Total: TAK-243 1 mg, 2 mg, 4 mg, 8 mg, 12 mg, 18 mg, and 4mg homozygous mutant, infusion, IV over 10-minutes, twice-weekly on Days 1, 4, 8, and 11 in a 21-day treatment cycle for a maximum of 12 cycles, or until symptomatic deterioration or PD or discontinuation of study for another reason, or until study is stopped.
Arm/Group | Schedule A: TAK-243 Total
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.88 (12.101)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 79.69 (16.829)
Body Surface Area [Mean (Standard Deviation); unit: square meter (m^2)] | 1.936 (0.2364)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 10 Day 41)
Population: The safety population included all participants who received at least 1 dose of TAK-243.
Measure: Number; unit: participants
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
participants
  TEAEs | 3 | 4 | 4 | 4 | 4 | 8 | 1
  SAEs | 1 | 1 | 2 | 2 | 1 | 4 | 0

2. Primary Outcome: Number of Participants With Laboratory Related TEAEs by System Organ Class (SOC)
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 10 Day 41)
Population: The safety population included all participants who received at least 1 dose of TAK-243.
Measure: Number; unit: participants
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
participants
  Metabolism and nutrition disorders | 1 | 1 | 1 | 3 | 1 | 4 | 1
  Blood and lymphatic system disorders | 1 | 1 | 1 | 2 | 0 | 4 | 0
  Investigations | 1 | 1 | 2 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Vital Sign Related TEAEs by Preferred Term (PT)
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 10 Day 41)
Population: The safety population included all participants who received at least 1 dose of TAK-243.
Measure: Number; unit: participants
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
participants
  Pyrexia | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Dyspnoea | 0 | 0 | 1 | 0 | 0 | 2 | 0
  Dyspnoea exertional | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypertension | 0 | 0 | 1 | 0 | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Time Frame: Cycle 1 Day 1 up to Cycle 1 Day 11
Population: The safety population included all participants who received at least 1 dose of TAK-243.
Measure: Number; unit: participants
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Echocardiogram Abnormalities
Time Frame: Cycle 1 Day 2 up to 30 days after last dose of study drug (Cycle 10 Day 41)
Population: The safety population included all participants who received at least 1 dose of TAK-243.
Measure: Number; unit: participants
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With TEAEs Related to Tropinin I and T
Time Frame: Baseline up to 30 days after last dose of study drug (Cycle 10 Day 41)
Population: The safety population included all participants who received at least 1 dose of TAK-243.
Measure: Number; unit: participants
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
participants | 0 | 0 | 1 | 0 | 0 | 0 | 0

7. Secondary Outcome: Ceoi: Plasma Concentration at the End of Infusion for TAK-243
Time Frame: Cycle 1 Day 1 and 11: pre-infusion to end of infusion (up to 10 minutes)
Population: The plasma pharmacokinetic (PK) analysis population where data at specified time points was available.The plasma PK-evaluable population included all participants who have sufficient dosing and concentration-time data to reliably estimate PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 8 | 1
  Cycle 1 Day 1 | 78.658 (48.2212) | 100.758 (24.0669) | 473.075 (132.7667) | 921.804 (258.6109) | 1276.684 (804.4476) | 1775.470 (463.8601) | 391.000 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.
  Cycle 1 Day 11: number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 7 | 1
  Cycle 1 Day 11 | 68.073 (35.2718) | 129.681 (52.4680) | 273.807 (179.4241) | 2299.438 (9027.7420) | 1271.199 (628.4555) | 2316.282 (7744.9842) | 265.000 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

8. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-243
Time Frame: Cycle 1 Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose; Cycle 1 Day 11 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The plasma PK analysis population where data at specified time points was available. The plasma PK-evaluable population included all participants who have sufficient dosing and concentration-time data to reliably estimate PK parameters.
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
nanogram hours per milliliter (ng*hr/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 5 | 0
  Cycle 1 Day 1 | 32.853 (17.3894) | 52.845 (5.6656) | 312.714 (193.3829) | 368.071 (8.2218) | 867.427 (374.1800) | 922.068 (192.2359) |
  Cycle 1 Day 11: number analyzed (Participants) | 3 | 4 | 1 | 0 | 0 | 0 | 1
  Cycle 1 Day 11 | 30.181 (12.8884) | 50.337 (8.9494) | 178.142 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  | 228.053 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis.

9. Secondary Outcome: AUCτ: Area Under the Plasma Concentration-time Curve Over the Dosing Interval for TAK-243
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 5 | 0
  Cycle 1 Day 1 |  |  | 535.581 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 377.812 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 1132.160 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 922.059 (192.1773) |
  Cycle 1 Day 11: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 5 | 0
  Cycle 1 Day 11 |  |  |  | 506.693 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 663.176 (261.1957) | 771.491 (181.7875) |

10. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-243
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
ng*hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 3 | 4 | 0
  Cycle 1 Day 1 |  |  | 203.043 (10.0600) | 375.541 (11.2872) | 579.122 (201.1755) | 768.728 (174.9927) |
  Cycle 1 Day 11: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 3 | 0
  Cycle 1 Day 11 |  |  | 179.726 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 509.785 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 752.152 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 864.533 (175.9351) |

11. Secondary Outcome: CL: Total Clearance After Intravenous Administration for TAK-243
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
liter per hour (L/hr)
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 3 | 4 | 0
  Cycle 1 Day 1 |  |  | 19.724 (0.9773) | 21.312 (0.6406) | 22.749 (8.8967) | 24.379 (5.6587) |
  Cycle 1 Day 11: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 3 | 0
  Cycle 1 Day 11 |  |  | 22.162 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 15.789 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 16.194 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 21.558 (4.8376) |

12. Secondary Outcome: Vss: Volume of Distribution at Steady State for TAK-243
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
liter
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 3 | 4 | 0
  Cycle 1 Day 1 |  |  | 29.806 (0.9494) | 33.957 (5.8273) | 37.596 (20.7520) | 63.744 (39.5945) |
  Cycle 1 Day 11: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 3 | 0
  Cycle 1 Day 11 |  |  | 34.120 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 39.618 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 56.573 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 51.806 (18.8787) |

13. Secondary Outcome: Aet: Amount of TAK-243 Excreted Unchanged in Urine
Time Frame: Cycle 1 Day 1; Cycle 1 Day 11
Population: No data were collected as no participant was analyzed since study was terminated before the planned expansion phase.
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Fet: Percentage of TAK-243 Excreted Unchanged in Urine
Time Frame: Cycle 1 Day 1; Cycle 1 Day 11
Population: No data were collected as no participant was analyzed since study was terminated before the planned expansion phase.
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for TAK-243
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 4 | 4 | 5 | 8 | 1
hour
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 2 | 2 | 3 | 4 | 0
  Cycle 1 Day 1 |  |  | 7.001 (1.4372) | 9.377 (4.6442) | 5.765 (0.8607) | 8.296 (4.3573) |
  Cycle 1 Day 11: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 3 | 0
  Cycle 1 Day 11 |  |  | 5.572 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 15.212 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 27.446 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 9.873 (6.3030) |

16. Secondary Outcome: Change From Baseline in Immunohistochemistry (IHC) Biomarkers in Tumor Biopsies at Cycle 1 Day 12 (C1D12) as Assessed by Histological Score (H-score)
Description: The pharmacodynamics IHC biomarkers included polyubiquitin marker and ubquityl (Ub)-histone H2B marker. H-score was a composite score that comprised of intensity and percentage of staining and was used for assessing the amount of protein or phospho-protein present in a biopsy sample. The composite score obtained by H-score is derived by summing the percentages of cell staining at each intensity multiplied by the weighted intensity of staining (0, 1+, 2+, 3+; where 3+ indicates the strongest staining, 2+ indicates medium staining, 1+ indicates weak staining, and 0 indicates no staining). The composite H-score ranges from 0 to 300, with a score of 0 representing the absence of any of the target protein and an H-score of 300 representing maximum staining and intensity of the target protein.
Time Frame: Baseline and Cycle 1 Day 12
Population: Pharmacodynamic population:baseline,post-baseline assessments were available,including all participants who received all doses(Cycle 1),have pre-post dose paired tumor tissue biopsies taken at protocol-specified timepoints,have sufficient tumor content at both timepoints to estimate changes in Pharmacodynamic biomarker percent area positive values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0 | 0
score on a scale
  Baseline: Polyubiquitin H-score | 286.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 297.80 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 282.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  |
  Change at C1D12: Polyubiquitin H-score | -3.60 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | -2.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 4.20 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  |
  Baseline: Ub-histone H2B H-score | 269.750 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 291.000 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 290.750 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  |
  Change at C1D12: Ub-histone H2B H-score | 13.250 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 3.250 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 2.000 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  |

17. Secondary Outcome: Change From Baseline in IHC Biomarkers in Tumor Biopsies at C1D12 as Assessed by Positive Index
Description: The pharmacodynamics IHC biomarkers included polyubiquitin marker and Ub-histone H2B marker. Positive index was calculated by taking the number of positive cells over the total number of cells.
Time Frame: Baseline and Cycle 1 Day 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: percentage of cell
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0 | 0
percentage of cell
  Baseline: Polyubiquitin Positive Index | 0.99 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 1.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.99 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  |
  Change at C1D12: Polyubiquitin Positive Index | -0.01 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.00 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  |
  Baseline: Ub-histone H2B Positive Index | 0.953 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.995 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.990 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  |
  Change at C1D12: Ub-histone H2B Positive Index | 0.018 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | 0.003 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. | -0.003 (NA) — Standard deviation could not be calculated since only 1 participant was available for analysis. |  |  |  |

18. Secondary Outcome: Percentage of Participants With Best Overall Response
Description: Best overall response for participant is best observed post-baseline disease response as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target and non target) must have reduction in short axis to less than (<) 10 millimeter (mm). Partial Response (PR): at least 30 percent (%) decrease in sum of diameter of target lesions, taking as reference baseline sum of diameter. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum of diameter; PD: at least 20% increase in sum of diameter of target lesions, taking as reference, smallest sum on study (this includes baseline sum if that is smallest on study). In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least mm. The appearance of 1 or more new lesions is also considered progression.
Time Frame: Baseline up to end of study (approximately 7 months)
Population: The response-evaluable population included all participants who received at least 1 dose of TAK-243, have measurable disease at baseline, and have at least 1 post baseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 3 | 4 | 2 | 3 | 2 | 5 | 1
percentage of participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 33 | 0 | 0 | 0 | 0 | 0 | 0
  SD | 67 | 75 | 100 | 0 | 50 | 60 | 0
  PD | 0 | 25 | 0 | 100 | 50 | 40 | 100

19. Secondary Outcome: Duration of Response
Description: Duration of any response (CR or PR) was defined as the time (in both days and months) from the date of first documented response per the investigator response assessment to the date of first progressive disease after the first documented response or, if the participant discontinues treatment, the date of last disease assessment as per RECIST version 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target and non target) must have reduction in short axis to <10 mm. PR: at least 30% decrease in sum of diameter of target lesions, taking as reference baseline sum of diameter.
Time Frame: Baseline up to end of study (approximately 7 months)
Population: The response-evaluable population where baseline and post-baseline assessments were available. The Response-evaluable population included all participants who received at least 1 dose of TAK-243, have measurable disease at baseline, and have at least 1 post baseline disease assessment.
Measure: Median (Full Range); unit: months
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0
months | 6.24 [6.24 to 6.24] |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days (Cycle 10 Day 41) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Schedule A: TAK-243 1 mg | Schedule A: TAK-243 2 mg | Schedule A: TAK-243 4 mg | Schedule A: TAK-243 8 mg | Schedule A: TAK-243 12 mg | Schedule A: TAK-243 18 mg | Schedule A: TAK-243 Homozygous Mutant 4 mg
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/4 | 2/4 | 2/4 | 1/5 | 4/8 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 4/4 | 4/4 | 3/5 | 8/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A: TAK-243 1 mg (N=3) | Schedule A: TAK-243 2 mg (N=4) | Schedule A: TAK-243 4 mg (N=4) | Schedule A: TAK-243 8 mg (N=4) | Schedule A: TAK-243 12 mg (N=5) | Schedule A: TAK-243 18 mg (N=8) | Schedule A: TAK-243 Homozygous Mutant 4 mg (N=1)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viraemia and fungaemia not elsewhere classified (NEC) (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenal and small intestinal stenosis and obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence, bloating and distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule A: TAK-243 1 mg (N=3) | Schedule A: TAK-243 2 mg (N=4) | Schedule A: TAK-243 4 mg (N=4) | Schedule A: TAK-243 8 mg (N=4) | Schedule A: TAK-243 12 mg (N=5) | Schedule A: TAK-243 18 mg (N=8) | Schedule A: TAK-243 Homozygous Mutant 4 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medical device site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical device site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Abscess oral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 (0) | 1 | 0
Troponin T increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.